CLINICAL TRIAL: NCT03705208
Title: Long-term Evaluation of the Effects of Youth First on Social and Emotional Development, Gender Equity, and Health of Adolescents in Rural Bihar, India
Brief Title: Youth First: A Longitudinal Impact Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CorStone (Other)
Collaborators: David and Lucile Packard Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01-YF-IN-2018-V1
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Resilience, Psychological; Mental Health Wellness 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Youth First Curriculum (Experimental): The full Youth First curriculum provides holistic training of both emotional resilience and adolescent health concepts. The curriculum is comprised of a 15-session emotional resilience curriculum and a 10-session adolescent health program. The resilience curriculum aims to increase both internal assets (such as self-esteem, coping skills, health knowledge, and conflict-resolution skills) and external assets (such as positive bonds with peers and family).
  The adolescent health curriculum provides in-depth training in physical health and wellness topics such as sexual and reproductive health, common diseases, nutrition, gender equality, and substance use.
  The curriculum is imparted by school teachers are trained and certified by CorStone.
  Interventions: Other: Youth First Curriculum
- School as usual (No Intervention): This arm is comprised of students attending school as usual and receiving the established government-designed curriculum.

INTERVENTIONS:
Other: Youth First Curriculum — A 25 session emotional resilience and health curriculum designed for 7th and 8th grade students.
  Other Names: School-based emotional resilience and health curriculum
  Arms: Youth First Curriculum

SUMMARY:
This trial will assess the effect of school-based emotional resilience and health curriculum, called Youth First, on middle school students who receive the curriculum in 7th and 8th grades. Key psychosocial wellbeing, mental health, educational wellbeing and substance use measures, will be assessed longitudinally over a three year period using a cluster randomized control design.

DETAILED DESCRIPTION:
This protocol is designed to answer key questions about the effects of Youth First on mental and sexual reproductive health, educational wellbeing and substance use. A mixed-methods, cluster randomized trial will assess the impact of the Youth First program over time. This component of the Youth First impact evaluation will take place across 70 schools (40 schools that are new to the Youth First intervention, 30 control schools) with 7th and 8th Standard students located within two districts in the state of Bihar, India, specifically Patna and Darbhanga.

This study will follow two cohorts of students: one of 8th Standard students and the other 7th Standard. This will include surveys conducted at baseline and at three follow-up time periods across a period of 32 months post-baseline (follow-up data collection at 8 (T1), 20 (T2), 32 (T3) months) to determine the short and long-term impact and additive effects of multiple years of Youth First. Eighth standard students will be followed through the end of 10th standard; the 7th standard cohort will be followed through the end of 9th. Both students who stay in school and those who leave will be followed up.

Quantitative data will be collected from 7th Standard (n=4500) and 8th Standard (n=3690) boys and girls across 100 schools in the two sub-studies, for a total study population of N=8190 students. Monitoring data from schools (e.g. number of sessions implemented, adherence to curriculum, etc.) collected as part of program implementation will inform a process evaluation of program quality and fidelity. Qualitative data will be collected from students after the completion of the Youth First program at the end of 8th Standard and at the end of T3.

Findings from this program are expected to provide much-needed evidence about the long-term effects of programs to address the psychosocial needs of youths in India, as well as information on the scalability of such a program within the school setting. It is expected that the findings from this study will be used by policy makers to inform decision making around the implementation of Youth First or similar programs within the state of Bihar and nationwide.

ELIGIBILITY:
Inclusion Criteria:

* All students enrolled in 7th or 8th grades at one of the schools selected for the study.

School Selection Criteria are:

* Government-run schools classified as rural and located in Darbhanga or Patna districts
* Have a minimum of 30 students enrolled in each of 7th and 8th Standards
* Have a high level of commitment from the principal to implement Youth First in both 7th and 8th grades, including willingness to have their teachers attend the training sessions and take the time to carry out the weekly sessions with the students.
* Have a high level commitment from the teachers of 7th and 8th Standards to participate in Youth First sessions, which includes taking part in all 3 trainings and holding weekly Youth First sessions.
* Have a physical space regularly available in which sessions could be held (relatively private and quiet, clean and uncluttered)
* Have a regular student teacher ratio of 50:1 or below (based on data reported in U-DISE)
* Accessible by a bus or taxi ride not greater than 3 hours from the nearest urban center.
* Classified as rural school by the Bihar Education Program Council

Exclusion Criteria:

* No exclusion criteria for students.

School exclusion criteria are:

* Have experienced a delay in starting the school year in AY2017/18.
* Have experienced extensive flooding in AY2017/18.
* Currently implementing a similar emotional resilience or life skills program in the middle school levels.
* Located in Naxal-affected area

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7762 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of student reporting being enrolled and regularly attending school | 32 months
  Participants are enrolled in a grade-appropriate school at the end of the study period
Substance use | 32 months
  Self-reported use of tobacco, alcohol or drugs.
Mental health | 32 months
  Strengths and Difficulties Questionnaire, internalizing problems subscale: Sum of 10 items, score range of 0-20, with lower score indicating better outcomes.
  KIDSCREEN psychological wellbeing: sum of 5 items, score range of 0-20 with higher score indicating better outcomes.
Physical Health | 32 months
  KIDSCREEN Physical wellbeing subscale: sum of 5 items, score range of 0-20 with higher score indicating better outcomes.

SECONDARY OUTCOMES:
Gender equitable attitudes | 8, 20 and 32 months
  Global Early Adolescent gender equity measure
Emotional Resilience | 8, 20 and 32 months
  Connor-Davidson Resilience measure: measure of emotional resilience. Sum of 10 items. Scale range from 0-40. Higher score indicates better outcomes.
Self-efficacy | 8, 20 and 32 months
  Schwarzer's Self-Efficacy Scale: Sum of 10 items. Scale range from 0-40. Higher score indicates better outcome.
Social Wellbeing | 8, 20 and 32 months
  KIDSCREEN Social Wellbeing: sum of 5 items, score range of 0-20 with higher score indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Elkins, PhD, Principal Investigator — CorStone
Locations (1):
- CorStone India Foundation, New Delhi, India

IPD SHARING:
Plan to Share IPD: No